CLINICAL TRIAL: NCT03620565
Title: A Multi-center Study: The Follow-up of Complications for Women Having Pelvic Reconstruction Surgery With Mesh/Native Tissue(Part I)
Brief Title: The Follow-up of Mesh/Native Tissue Complications Study(Part I)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Peking University People's Hospital (Other); Qilu Hospital of Shandong University (Other); Obstetrics & Gynecology Hospital of Fudan University，Shanghai Red House Obstetrics & Gynecology Hospital (Unknown); Peking University Third Hospital (Other); First Hospitals affiliated to the China PLA General Hospital (Other Government); Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other); Tongji Hospital (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Wuxi Obsetrics & Gynecology Hospital (Unknown); Fuzhou General Hospital (Other); The First Affiliated Hospital of Jinan Hospital (Unknown); Women's Hospital School Of Medicine Zhejiang University (Other); Renmin Hospital of Wuhan University (Other); The Third Hospital Affiliated Zhengzhou University (Unknown); Shengjing Hospital (Other); General Hospital of Ningxia Medical University (Other); The Second Hospital of Hebei Medical University (Other); Gansu Provincial Maternal and Child Health Care Hospital (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Yantai Yuhuangding Hospital，Medical College, Qingdao University (Unknown); Southwest Hospital, China (Other); West China Second University Hospital (Other); Jiangxi Maternal and Child Health Hospital (Other); Shanxi Coal Central Hospital (Unknown); Chongqing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: JS-1566-1
Record Dates: First submitted 2018-07-06; First posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-06

CONDITIONS: Pelvic Floor
Keywords: Pelvic floor reconstructive surgery; Mesh; Native tissue; Tape; Complication; the CTS coding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Laparoscopic sacrocolpopexy(LSC): Patients who prefer to accept laparoscopic sacrocolpopexy after hysterectomy. For patients who has desire of uterine-preservation,laparoscopic sacrocervicopexy or sacrohysteropexy is carried.
- Reconstruction with transvaginal mesh(TVM): Patients who undertake pelvic reconstruction with tran-vaginal mesh(commercial mesh kits or self-cut synthesized mesh).
- Reconstruction with native tissue(NT): Patients who prefer to accept reconstruction with native tissue,mainly including high uterosacral ligament suspension, sacrospinous ligament fixation,ischial spinous fascia fixation,the Lefort operation.
- Tension-free vaginal tape surgery(TVT): Patients who undertake anti-incontinence surgeries(tension-free vaginal tape procedure).

SUMMARY:
This study aims to investigate the incidence and distribution of complications after different pelvic reconstruction surgeries using mesh/native tissue in multi-centers using the IUGA/ICS complication classification system(the Category-Time-Site(CTS) coding).

DETAILED DESCRIPTION:
Patients who undergo different pelvic floor reconstructive surgeries for the cure of pelvic organ prolapse(POP)and/or stress urinary incontinence(SUI) between June 2018 and June 2023 from 27 tertiary hospitals are prospectively collected.Our study aims to follow-up and report the incidences of postoperative complications according to the International Urogynecological Association-International Continence Society(IUGA-ICS) Complication Classification Coding(Category-Time-Site coding system).The aimed pelvic floor reconstructive surgeries involve anterior,apical, posterior or total pelvic reconstruction with trans-vaginal mesh,open/laparoscopic sacrocolpopexy(Y-tape/self-cut synthesized mesh),repair using native tissue(sacrospinous ligament fixation, high uterosacral ligament suspension,ischial spinous fascia fixation, the Lefort operation and so on)and as well as anti-urinary incontinence surgeries(tension-free vaginal tape).

Our follow-up process start after patients have completed the operation,thus our study do not affect patients' choice of surgical method.

ELIGIBILITY:
Inclusion Criteria:

- 1. Patients who undergo pelvic floor reconstructive surgeries for pelvic organ prolapse and/or stress urinary incontinence. The aimed pelvic floor reconstructive surgeries involve anterior, apical, posterior or total pelvic reconstruction with trans-vaginal mesh, open/laparoscopic sacrocolpopexy (Y-shape tape/self-cut synthesized mesh), repair using native tissue(sacrospinous ligament fixation, high uterosacral ligament suspension, ischial spinous fascia fixation, the Lefort operation and so on) and as well as anti-urinary incontinence surgeries(tension-free vaginal tape). The indications are respectively as follows:

1. Total pelvic reconstruction with trans-vaginal mesh Indications: 1) Patients experienced recurrence of prolapse in the same compartment that has a history of pelvic floor repair surgery; 2) The choice for elder patients who will accept primary surgery for advanced POP (staging III or IV).
2. Open/Laparoscopic sacrocolpopexy (Y-shape tape/self-cut synthesized mesh) Indications: 1) Presenting with at least 3 prolapse of the uterus, with or without concomitant cystocele and rectocele; 2) Symptomatic stage 2 or greater prolapse of the vaginal vault or apical recurrence.
3. Repair using native tissue(sacrospinous ligament fixation, high uterosacral ligament suspension, ischial spinous fascia fixation, Lefort) Indications:1)Presenting symptomatic stage 2 or greater prolapse of the uterus, with or without concomitant cystocele and rectocele. The procedure(sacrospinous ligament fixation, high uterosacral ligament suspension, ischial spinous fascia fixation) usually is performed after hysterectomy or when the uterus is preserved. 2)If postmenopausal women present with advanced uterus or vaginal apex prolapse, and have no desire of sexual life, the Lefort operation would be performed.
4. Anti-urinary incontinence surgeries: tension-free vaginal tape. Indications: Stress urinary incontinence(SUI) patients who have 1）hyperactivity of urethra, or 2）internal urethral sphincter disorder; Or 3）mainly presenting SUI symptoms in patients with mixed urinary incontinence.

2. The failure or recurrence of prolapse the same compartment that has been underwent repair using native tissue.

Exclusion Criteria:

* (1) the recurrence occurred on the same pelvic compartment with a prior history of prolapse repair surgery using mesh, an implant or a graft; (2) a prior history of anti-incontinence surgery using tape; however, patients who are inferred to accept procedures for POP this time are not included; (3) acute/chronic pelvic inflammation, genital tract infections；(4) any severe medical diseases that precluded the operations.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who undergo different pelvic floor reconstructive surgeries for the cure of pelvic organ prolapse (POP) and/or stress urinary incontinence (SUI) between June 2018 and June 2023 from 27 tertiary hospitals are prospectively collected.
Sampling Method: Non-Probability Sample
Enrollment: 13120 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The frequency and incidence rate of different complications | at 6-week postoperatively
  Postoperative follow-up and record the occurrence of complications according to the International Urogynecological Association-International Continence Society（IUGA-ICS）Complication Classification Coding(Category-Time-Site coding system).
The frequency and incidence rate of different complications | at 3-month postoperatively
  Postoperative follow-up and record the occurrence of complications according to the International Urogynecological Association-International Continence Society（IUGA-ICS）Complication Classification Coding(Category-Time-Site coding system).
The frequency and incidence rate of different complications | at 1-year postoperatively
  Postoperative follow-up and record the occurrence of complications according to the International Urogynecological Association-International Continence Society（IUGA-ICS）Complication Classification Coding(Category-Time-Site coding system).
The frequency and incidence rate of different complications | at 2-year postoperatively
  Postoperative follow-up and record the occurrence of complications according to the International Urogynecological Association-International Continence Society（IUGA-ICS）Complication Classification Coding(Category-Time-Site coding system).
The frequency and incidence rate of different complications | up to 3-year postoperatively
  Postoperative follow-up and record the occurrence of complications according to the International Urogynecological Association-International Continence Society（IUGA-ICS）Complication Classification Coding(Category-Time-Site coding system).

SECONDARY OUTCOMES:
Anatomical cure rates in treated compartment of different pelvic reconstructive surgeries | 6 weeks, 3 months and each year, up to 3-year postoperatively
  The percentage of patients who reach the anatomical success criteria at each time point（6 weeks, 3 months and each year, up to 3-year postoperatively）
Change from Preoperative scores of POP-Q(Pelvic organ prolapse quantitation) at each follow-up | Preoperatively; At 6weeks, 3 months, 1 year and assessed up to 3 year postoperatively.
  POP-Q is used for evaluation the severity(staging) of prolapse by pelvic examination preoperatively and postoperatively. The score is reported in cm. The changes from baseline scores at 6 weeks, 3 months, 1 year and up to 3 years postoperatively are respectively compared.

CONTACTS AND LOCATIONS:
Overall Officials: Lan Zhu, MD, Principal Investigator — Peking Union Medical College Hospital, Chinese Academy of Medicine Sciences
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medicine Sciences, Beijing, Beiing, China

REFERENCES:
- [Derived] Sun ZJ, Wang XQ, Lang JH, Xu T, Lu YX, Hua KQ, Han JS, Li HF, Tong XW, Wang P, Wang JL, Yang X, Huang XH, Liu PS, Song YF, Jin HM, Xie JY, Wang LW, Wu QK, Gong J, Wang Y, Wang LQ, Li ZA, Xu HC, Xia ZJ, Gu LN, Liu Q, Zhu L. A 14-year multi-institutional collaborative study of Chinese pelvic floor surgical procedures related to pelvic organ prolapse. Chin Med J (Engl). 2021 Jan 20;134(2):200-205. doi: 10.1097/CM9.0000000000001237. PMID 33443938